CLINICAL TRIAL: NCT06358235
Title: Evaluation of The Effect of Music Therapy on Dyspnea Severity and Vital Signs In Intensive Care Patients
Brief Title: The Effect of Music Therapy on Dyspnea Severity and Vital Signs
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, Hafize Aydemir, Principal Investigator, Suleyman Demirel University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SDU-IH-HA-01
Record Dates: First submitted 2024-04-02; First posted 2024-04-10 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Dyspnea; Chronic Obstructive Pulmonary Disease
Keywords: Music Therapy; Dyspnea; İntensive Care; Vital Signs
MeSH Terms: conditions — Dyspnea; Pulmonary Disease, Chronic Obstructive | interventions — Music Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music Therapy (Experimental): The Patient Identification Form, Modified Borg Scale, Vital Signs Record Chart, and Blood Test Results Record Chart will be completed when the patient is first admitted to the ward. Music therapy intervention will be administered between 6:00 AM and 12:00 PM. Before the music therapy session, the patient will lie on their back at a 30-45 degree angle and rest for 5 minutes. The Modified Borg Scale and Vital Signs Record Chart will be completed just before the music therapy session begins. During the session, the patient will receive the music therapy intervention through headphones for 30 minutes. At the end of the 30-minute music session, the Modified Borg Scale and Vital Signs Record Chart will be completed again. Thirty minutes after the end of the music therapy intervention, the Modified Borg Scale and Vital Signs Record Chart will be completed once more.
  Interventions: Other: Music Therapy
- No Music Therapy (Other): When the patient is admitted to the ward, the Patient Identification Form, Modified Borg Scale, Vital Signs Record Chart, and Blood Test Results Record Chart will be completed. Music therapy will not be applied to this group; however, patients will be provided with headphones to maintain consistent conditions. When the patient is ready, between 6:00 AM and 12:00 PM, they will lie on their back at a 30-45 degree angle and rest for 5 minutes. The Modified Borg Scale and Vital Signs Record Chart will be completed just before the patient puts on the headphones. Once the session begins, the patient will quietly spend 30 minutes with headphones. After 30 minutes, the Modified Borg Scale and Vital Signs Record Chart will be filled out again. Thirty minutes after the end of the session, the Modified Borg Scale and Vital Signs Record Chart will be completed again.
  Interventions: Other: No Music therapy

INTERVENTIONS:
Other: Music Therapy — 30-minute music therapy session.
  Arms: Music Therapy
Other: No Music therapy — The practice where patients are simply fitted with headphones and rest quietly without listening to music.
  Arms: No Music Therapy

SUMMARY:
This study aims to investigate the effect of music therapy on dyspnea severity and quality of life indicators in patients with Chronic Obstructive Pulmonary Disease (COPD) admitted to the intensive care unit. The study will be conducted at Isparta City Hospital and Kumluca State Hospital in Antalya, Turkey, using an experimental design. Patients will be divided into experimental and control groups, selected using randomization.

Patients in the experimental group will receive music therapy in the Hüseyni maqam, while those in the control group will not receive any music therapy. Life indicators and Modified Borg Scale (MBS) values of patients in the experimental group will be recorded before, immediately after, and 30 minutes post-application. Music therapy will be administered to patients for only one day, once in the morning. Data for patients in the control group will be collected at the same time intervals. The results of this study aim to contribute to the literature on the impact of music therapy on dyspnea severity and quality of life indicators in COPD patients.

DETAILED DESCRIPTION:
Intensive care is a multidisciplinary, professional field where patients with acute, life-threatening conditions or at risk of organ dysfunction are comprehensively managed. The primary goal of intensive care is to treat existing physical problems while maintaining the patient's physiological course and preventing deterioration. Perceiving breathing as strenuous and abnormal is defined as dyspnea. Assessing the severity of dyspnea is an important indicator for the progression of the disease. Dyspnea affects an individual's daily life, negatively impacting their ability to perform physical activities . Music therapy, as part of medical care, can be effectively used in the treatment of lung diseases and symptoms. It is enjoyable, cost-effective, and applicable almost anywhere . Music is reported to be effective as a pharmacological and non-invasive intervention in alleviating breathlessness .

The psychological and physical effects of music on humans have long been recognized. Music, by following a specific physiological pathway, can have various effects on the body, from reducing anxiety to lowering blood pressure and inducing relaxation. It is believed that negative thoughts and experiences can lead to physiological and psychological illness. Music is believed to have a profound impact on these illnesses .

There are limited studies in our country that investigate the effects of music therapy on patients admitted to intensive care with dyspnea complaints. In conclusion, dyspnea is a common problem among patients admitted to intensive care with a diagnosis of COPD. This study is planned to evaluate how music therapy affects dyspnea severity and life indicators in COPD patients admitted to intensive care. It is believed that the findings will contribute to the literature in terms of nursing care.

ELIGIBILITY:
Inclusion Criteria:

* Being treated as a patient in intensive care.
* Being monitored with a diagnosis of COPD (Chronic Obstructive Pulmonary Disease).
* Currently undergoing treatment for dyspnea symptoms.
* Volunteering to participate in the research.
* Receiving treatment at Kumluca State Hospital.
* Receiving treatment at Isparta City Hospital.
* Being 18 years of age or older.
* Having intact consciousness and full capacity for judgment.
* Being able to read and write.
* Speaking Turkish.
* Having no communication barriers.

Exclusion Criteria:

* Decline participation in the research.
* Wish to withdraw from the study after it has started.
* Have a verbal communication barrier.
* Be under 18 years of age.
* Be receiving treatment in a unit other than intensive care.
* Have ear trauma, infection, or other ear-related conditions.
* Have hearing impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-01-07 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Patient Identification Form | Saving of values within 1 day. Evaluation of the data will take place within 3 months after the end of the study.
  The researcher has created a 12-question survey to determine patients' socio-demographic characteristics and health/medical history.
Modified Borg Scale | Saving of values within 2 day. Evaluation of the data will take place within 3 months after the end of the study.
  The Modified Borg Scale was initially developed by Borg in 1970. This scale was originally designed as a 6 to 20 rating scale to measure effort during physical activity. However, it was later modified into a 10-point system, including written indicators of severity. The Modified Borg Scale allows for the measurement of the severity of dyspnea (shortness of breath) in both resting and exertional states. It consists of a total of 10 items and enables patients to grade the severity of their dyspnea. Ratings are made on a scale from 0 to 10, where an increase in the number indicates an increase in dyspnea severity.
  The availability and comprehensibility of this scale make it quite easy to administer to patients. Moreover, its superiority over other scales measuring dyspnea severity has been proven in long-term use. Implementing the Modified Borg Scale as a significant component of your research will help us objectively evaluate changes in patients' dyspnea severity.
Vital Signs Record Chart | Saving of values within 2 day. Evaluation of the data will take place within 3 months after the end of the study.
  The chart was created by the researcher for recording the patient's blood pressure, pulse rate, respiratory rate, and saturation values.
Blood Test Results Record Chart | Saving of values within 1 day. Evaluation of the data will take place within 3 months after the end of the study.
  The chart was created by the researcher for recording the patient's blood test results.

CONTACTS AND LOCATIONS:
Locations (1):
- Suleyman Demırel University, Isparta, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No